CLINICAL TRIAL: NCT06128824
Title: High Frequency Imaging in Patients With Cerebral Amyloid Angiopathy
Brief Title: High Frequency Imaging in Cerebral Amyloid Angiopathy
Acronym: HIFI-CAA
Status: Active, not recruiting | Type: Observational
Sponsor: Martin Dichgans (Other)
Responsible Party: Sponsor-Investigator, Martin Dichgans, Director, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: HIFI-CAA-01
Record Dates: First submitted 2023-10-26; First posted 2023-11-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Amyloid Angiopathy
Keywords: cortical superficial siderosis; DWI+ lesion; serial imaging; disease progression; MRI; cerebrovascular events; focal subarachnoid hemorrhage
MeSH Terms: conditions — Cerebral Amyloid Angiopathy; Disease Progression | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with probable CAA and cSS or fSAH: Patients with probable CAA and cortical superficial siderosis (cSS) or focal subarachnoid haemorrhage (fSAH)
  Interventions: Other: MR Imaging
- Patients with probable CAA without cSS or fSAH: Patients with probable CAA and intracerebral hemorrhage (ICH; micro- or macrohemorrhage) but without cSS or fSAH
  Interventions: Other: MR Imaging

INTERVENTIONS:
Other: MR Imaging — Serial magnetic resonance imaging (MRI)

SUMMARY:
Cerebral amyloid angiopathy (CAA), caused by amyloid beta depositions in the walls of small cerebral vessels, is remarkably common in the elderly. Its major clinical consequences include intracerebral hemorrhages (ICH) typically in lobar location, functional dependence (disability) and cognitive impairment.

Cortical superficial siderosis (cSS) is a common finding in CAA patients and can even be the only magnetic resonance imaging sign of CAA. cSS is of high prognostic relevance regarding future intracerebral haemorrhage and disability. Previous studies suggest that cSS is caused by recurrent focal subarachnoid hemorrhages (fSAH). However, the exact mechanisms and the temporal dynamics of this highly relevant imaging finding are largely unknown.

In addition to hemorrhagic manifestations, such as cSS, CAA patients also show ischemic lesions. Of particular interest are acute ischemic lesions as detected by diffusion imaging, which seem to be highly prevalent. Since haemorrhagic and ischemic lesions require fundamentally different therapeutic strategies, understanding the relevance and interplay of both lesion types is highly important for clinical decision making.

The HIFI-CAA cohort study aims to provide novel insights into cSS, acute ischemic lesions and other relevant brain alterations in CAA through high-frequency (monthly) serial magnetic resonance imaging.

DETAILED DESCRIPTION:
Cerebral amyloid angiopathy (CAA) is defined as the deposition of β-amyloid in the walls of small cortical cerebral vessels. It is very common in the elderly population with prevalence rates up to 60% and is associated with Alzheimer´s disease. Intracerebral lobar macrohemorrhages (ICH) are the most devastating presentation of CAA and the main cause of morbidity and mortality. In addition to developing clinically manifest strokes, CAA patients may also suffer from transient neurological symptoms and progressive cognitive impairment ultimately resulting in dementia.

Apart from ICH, typical MRI signs of CAA include multiple cerebral microbleeds (CMB) in a cortical-subcortical localization, white matter hyperintensities on T2-weighted images and supratentorial cortical superficial siderosis (cSS). Main risk factors for recurrence of CAA-related ICH are apolipoprotein E ε2 or ε4 alleles, previous ICHs and CMB on follow-up imaging. Recently, cSS emerged as an additional, major independent risk factor for ICH and disability.

In CAA, siderosis affects the convexity of the cerebral hemispheres, and thus is termed cortical superficial siderosis (cSS). This is in contrast to infratentorial superficial siderosis, which is not linked to CAA. CSS is likely caused by recurrent non-traumatic, focal convexity subarachnoid hemorrhages (fSAH). There are causes of fSAH and cSS other than CAA, and these causes seem to vary depending on age: in younger patients (< 60 years of age) fSAH and cSS are most commonly seen in the context of trauma, vasculitis and reversible cerebral vasoconstriction syndrome, while CAA seems to be the by far most common cause in subjects above 60 years of age. cSS is common (> 60%) in patients with histologically proven CAA, and may be the only hemorrhagic imaging sign on MRI.

Lesions on diffusion-weighted imaging, i.e. areas of restricted diffusion, are a very frequent finding in CAA. These diffusion restrictions can be found in 25% to 50% of CAA patients when performing a single MRI. One recent study even suggests a spatial relationship with cSS. The clinical significance of these lesions is not yet fully established. The most likely pathophysiology behind these lesions is acute ischemia, or to be more precise cytotoxic edema after brain ischemia/infarction. However, subcortical infarcts as detected through a diffusion-restricted lesion can have vastly different fates, ranging from disappearance to complete brain tissue loss (cavitation). An important step in the understanding of these lesions is the precise estimation of prevalence and tissue consequences. A critical point in this endeavour is that these diffusion restricted lesions are typically only visible for a few weeks. Thus, they can remain completely undetected in studies using conventional study designs with follow-up intervals as long as 6 months, one year or even longer.

While small subcortical and cortical ischemic lesions (detectable as diffusion restrictions) are a common finding in CAA patients, their exact prevalence and relevance for disease progression are unclear. Overall, temporal dynamics of the processes leading to hemorrhagic and ischemic manifestations of CAA as well as their interrelationships are insufficiently understood. These critical aspects can be addressed by a novel study design with serial, monthly magnetic resonance imaging. The study design is inspired by a recent high-frequency serial imaging study in patients with sporadic, non-amyloid cerebral small vessel disease conducted at Nijmegen (Radboud University Nijmegen Diffusion tensor and Magnetic resonance imaging Cohort - Investigating The origin and Evolution of cerebral small vessel disease, RUN DMC - InTENse).

The primary aim of this study is to prospectively evaluate the development and temporal evolution of incident and prevalent fSAH & cSS in CAA patients.

Secondary aims are i) to assess the monthly incidence of acute ischemic lesions (diffusion restrictions) in CAA patients with cSS/fSAH and to compare the incidence with lobar ICH survivors, and ii) to assess the inter-relationship between hemorrhagic lesions (fSAH/cSS/CMB) and acute ischemic lesions as well as the association between these lesions and cerebrovascular event rates and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Probable CAA according to the modified Boston criteria with evidence of

  1. cSS or fSAH
  2. lobar ICH survivors without cSS or fSAH
* Absence of ICH or microbleed in deep locations (basal ganglia, thalamus, brain stem)
* Absence of infratentorial siderosis or infratentorial SAH
* MR-/CT-/DS-angiography without evidence of cerebral aneurysm, AVM, AV-fistula or other possible etiology for the observed haemorrhagic manifestations
* No history of head trauma resulting in loss of consciousness or radiologically visible traumatic brain injury
* Written informed consent by patient herself/himself prior to study enrolment

Exclusion Criteria:

* Unwillingness to participate in high-frequency (monthly) follow-up
* Severe medical condition with expected life expectancy <1 year
* Contraindications for MRI (following local guidelines of the respective study center)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be performed in a hospital-based setting. Patients with probable CAA according to the modified Boston criteria or Boston criteria v2.0 will be further evaluated for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
new hemorrhagic features as determined by heme-sensitive MRI | monthly up to 12 months
  new hemorrhagic features (e.g., cSS) as determined by heme-sensitive magnetic resonance imaging such as T2*-weighted gradient echo (GRE) and susceptibility weighted imaging (SWI)

SECONDARY OUTCOMES:
DWI+ lesions on diffusion weighted imaging MRI | monthly up to 12 months
  DWI+ lesions on diffusion weighted imaging (DWI) on magnetic resonance imaging
modified Rankin Scale | monthly up to 12 months
  functional outcome on modified Rankin Scale (score [0-6] with higher scores meaning a worse outcome)
neuropsychological evaluation (global cognition using MoCA) | baseline and after 12 months
  neuropsychological evaluation of cognition using the Montreal Cognitive Assessment (MoCA) (score [0-30] with higher scores meaning a better outcome)
neuropsychological evaluation (global cognition using MMSE) | baseline and after 12 months
  neuropsychological evaluation of cognition using the Mini Mental State Examination (MMSE) (score [0-30] with higher scores meaning a better outcome)
neuropsychological evaluation (processing speed and executive function) | baseline and after 12 months
  neuropsychological evaluation of processing speed and executive function using the Trail Making Test (TMT) A and TMT B measuring the time in seconds to complete the task; age- and education-corrected z-scores will be derived
reaction time (attention) | monthly up to 12 months
  reaction time assessed with Test of Attentional Performance (TAP) test

CONTACTS AND LOCATIONS:
Overall Officials: Marco Duering, MD, Principal Investigator — Institute for Stroke and Dementia Research
Locations (3):
- Germany (3):
  - DZNE/Bonn - Klinik und Poliklinik für Neurologie, Universitätsklinikum Bonn, Bonn
  - DZNE/Magdeburg - Universitätsklinikum Magdeburg, Magdeburg
  - Insitute for Stroke and Dementia Research, Munich

IPD SHARING:
Plan to Share IPD: Undecided
has to be further decided, upon reasonable request